CLINICAL TRIAL: NCT02114307
Title: REVITIVE for the Treatment of Patients With Venous Insufficiency
Acronym: RVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Actegy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13HH0768
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Results first posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-09

CONDITIONS: Venous Insufficiency; Oedema; Varicose Veins
Keywords: electrical stimulation; venous insufficiency; post thrombotic syndrome; varicose veins
MeSH Terms: conditions — Venous Insufficiency; Edema; Varicose Veins; Postthrombotic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REVITIVE IX: actual device (Active Comparator): Trial participants will receive the true Revitive IX device
  Interventions: Device: REVITIVE IX
- REVITIVE IX: sham device (Sham Comparator): Trial participants will receive a sham device
  Interventions: Device: REVITIVE IX

INTERVENTIONS:
Device: REVITIVE IX — neuromuscular electrical stimulation device

SUMMARY:
To investigate the efficacy of an electrical stimulation (using the REVITIVE IX device) in treating patients with venous insufficiency.

DETAILED DESCRIPTION:
This is a pilot randomised control trial to assess the efficacy of a neuromuscular electrical stimulation device to improve venous blood flow and patients' symptoms in patients with chronic venous insufficiency. The Revitive IX device is a neuromuscular electrical stimulation device that gives wide pulse pattern electrical stimulation via foot pads. A cycle of treatment consists of a 30 minute programme of 15 varying waveforms that last a minute each.

Twenty patients with venous insufficiency will be screened according the eligibility criteria. Patients will be randomised to either treatment or control (sham device) group. Patients are advised to use the device 30 minutes a day, everyday, for 6 weeks. Compliance will be monitored with a data logger and diary card.

Primary outcome measure:

a) improvement in venous haemodynamics.

Secondary outcome measures:

1. improvement in lower limb oedema
2. improvement in clinical symptoms
3. reduction in lower limb pain and discomfort
4. improvement in quality of life measures
5. device satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study and provide meaningful written informed consent for the study.
* Willing, able, and committed to participate in the procedures for the full length of the study.
* All ethnic groups, male or female above the age of 18 years.
* Diagnosis of chronic venous insufficiency (C2-C5 CEAP classified)
* Be of non-childbearing potential; or using adequate contraception and have a negative urine pregnancy test result within 24 hours if appropriate before using the device.
* Blood pressure currently under moderate control (<160/100mmHg)
* No current foot ulceration.

Exclusion Criteria:

* Has insufficient ability to understand the subject information sheet, consent form and verbal instruction.
* Has an unstable condition (eg psychiatric disorder, a recent history of substance abuse or otherwise thought to be unreliable or incapable of complying wight he requirements of the clinical investigational plan (CIP).
* Has any metal implants.
* Pregnant.
* Has a cardiac pacemaker, AICD or other implanted electrical device.
* Has an existing DVT.
* Has an acute medical condition other than chronic venous insufficiency.
* Has recent lower limb injury or lower back pain.
* Has current foot ulceration or other skin ulcers.
* Has cardiovascular disease.
* Has foot deformities.
* Has any disorder that, in the opinion of the investigator, might interfere with the conduct of the study.
* Has an ABPI < 0.8.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun Davies, MA DM FRCS FHEA, Principal Investigator — Imperial College London and Imperial College London NHS Trust
Locations (1):
- Academic Department of Vascular Surgery, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data available on request.
Supporting Information: Study Protocol, CSR
Time Frame: 12 Months after publication of main study
Access Criteria: From listed authors.

REFERENCES:
- [Result] Ravikumar R, Williams KJ, Babber A, Lane TRA, Moore HM, Davies AH. Randomised Controlled Trial: Potential Benefit of a Footplate Neuromuscular Electrical Stimulation Device in Patients with Chronic Venous Disease. Eur J Vasc Endovasc Surg. 2017 Jan;53(1):114-121. doi: 10.1016/j.ejvs.2016.09.015. Epub 2016 Dec 2. PMID 27919609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from vascular outpatients clinic between 20/02/2014 - 18/09/2014.
Pre-assignment Details: Patient stayed in the full length of the study. Chronic venous insufficiency (C2-C5 CEAP). Blood pressure <160/100mmHg. No current foot ulceration
Groups:
- REVITIVE IX: Sham Device: Trial participants will receive a sham device
  REVITIVE IX: sham device
Period: Overall Study
Arm/Group | REVITIVE IX: Actual Device | REVITIVE IX: Sham Device
Started | 11 | 11
Completed | 10 | 11
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test Device: Patients received the REVITIVE IX device for 6 weeks of home usage.
- Sham Device: Sham REVITIVE IX for 6 weeks of home usage.
- Total: Total of all reporting groups
Arm/Group | Test Device | Sham Device | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (12.4) | 54.6 (13.7) | 62.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Venous Haemodynamics - Percent Change in Time Averaged Mean Velocity TAMV
Description: Femoral vein haemodynamics is measured using ultrasound scan - Time Averaged Mean Velocity
Time Frame: 0 and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | REVITIVE IX: Actual Device | REVITIVE IX: Sham Device
Number analyzed (Participants) | 10 | 11
percentage change | 102.4 (50) | -9.1 (50)
Statistical Analysis 1: Comparison: REVITIVE IX: Actual Device vs REVITIVE IX: Sham Device; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Changes in Limb Swelling, Volume
Description: Lower limb oedema measured before and after using the device at 0 and 6 weeks using a perimeter.
  Limb volume was measured using an optoelectronic limb volumeter. Patients using compression stockings were advised to remove stockings 2 h prior to their appointment. Measurements were taken with the patient seated and the affected leg in a horizontal position. Five readings were taken before and after device usage at Week 0 and Week 6
Time Frame: 0 and 6 weeks
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Test Device | Sham Device
Number analyzed (Participants) | 10 | 11
ml
  week 0 prestimulation | 5377 (1122) | 5107 (1252)
  week 0 poststimulation | 5422 (1127) | 5208 (1252)
  week 6 prestimulation | 5500 (1173) | 5143 (1269)
  week 6 post stimulation | 5553 (1168) | 5203 (1272)
Statistical Analysis 1: Comparison: Sham Device; Sham Group - 6 week Time Point - Pre-stimulation versus Post-Stimulation; Test type: Superiority; p = 0.0023, t-test, 2 sided
Statistical Analysis 2: Comparison: Test Device; Test Group - 6 week Time Point - Pre-stimulation versus Post-Stimulation; Test type: Superiority; p = 0.0815, t-test, 2 sided

3. Secondary Outcome: Clinical Symptoms
Description: Change in clinical symptoms as assessed by the Venous Clinical Severity Score (VCSS) from 0 to 6 weeks, lower score means improvement. Maximum score on VCSS is 30. Minimum score is 0.
Time Frame: 0 and 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage change in VCSS score
Arm/Group | REVITIVE IX: Actual Device | REVITIVE IX: Sham Device
Number analyzed (Participants) | 11 | 10
Percentage change in VCSS score | -11.8 (31.2) | 6.4 (20.7)
Statistical Analysis 1: Comparison: REVITIVE IX: Actual Device vs REVITIVE IX: Sham Device; Test type: Superiority; p = 0.127, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | REVITIVE IX: Actual Device | REVITIVE IX: Sham Device
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes